CLINICAL TRIAL: NCT03403985
Title: Long-term Evaluation of Direct Pulp Capping Using Either Mineral Trioxid Aggregate or Calcium Hydroxide in Permanent Mature Teeth: A Randomized Controlled Trial
Brief Title: Long-term Evaluation of Direct Pulp Capping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JordanUST2
Record Dates: First submitted 2018-01-05; First posted 2018-01-19 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Dental Pulp Capping; Dental Caries Extending to Pulp
MeSH Terms: interventions — Calcium Hydroxide; mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Retrospective clinical trial
Who Masked: Participant
Masking Description: patients are not aware about type of capping material used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium hydroxide direct pulp capping (Experimental): calcium hydroxide (Ca(OH)2 direct pulp capping will be performed in this group
  Interventions: Drug: Calcium Hydroxide (Ca(OH)2)
- MTA direct pulp capping (Experimental): Mineral Trioxide Aggregate (MTA) direct pulp capping will be performed in this group
  Interventions: Drug: Mineral Trioxide Aggregate

INTERVENTIONS:
Drug: Calcium Hydroxide (Ca(OH)2) — Ca(OH)2 will be used in this group
  Other Names: Ca(OH)2
  Arms: calcium hydroxide direct pulp capping
Drug: Mineral Trioxide Aggregate — MTA will be used in this group
  Other Names: MTA
  Arms: MTA direct pulp capping

SUMMARY:
Calcium hydroxide and mineral trioxide aggregate have been used in vital pulp therapy with variable outcomes recorded by different study. They will be compared when used for direct pulp capping in cariously exposed mature permanent teeth.

DETAILED DESCRIPTION:
Vital pulp therapy has the benefit of providing patients with a conservative treatment option with relatively low cost when compared to conventional root canal treatment and spares them possible post-treatment consequences that might occur. Vital pulp treatment in trauma cases is associated with high success rate but controversy still exists regarding vital pulp treatment in carious-exposed pulp.

The purpose of this study is to evaluate the success rate of direct pulp capping performed with MTA-Angelus® or calcium hydroxide in mechanical-exposed or carious-exposed mature permanent human teeth. Patients included in this study will be recruited from routine dental patients attending conservative clinics in JUST Dental Teaching Centre. Adult patients scheduled for routine conservative treatment involving caries removal and restoration with mechanical or carious pulp exposure will be invited to participate in this study.

A total of 80 carious human teeth with carious pulp exposure will be included in this randomized clinical study. Patients are among those scheduled for conservative dental treatment and end with pulp exposure. The patients and/or their parents will be asked to sign a consent form after receiving a detailed explanation about the study rationale, clinical procedures, and possible risks. The exposed teeth will be divided randomly into two experimental groups (n=40) according to the dressing materials; MTA-Angelus® or calcium hydroxide, then teeth will be restored with permanent filling. Teeth will be reviewed recording any signs and symptoms. Patients will be reviewed in 1 week, 3 months and yearly after. MTA-Angelus and calcium hydroxide are anticipated to be biocompatible and induce hard tissue barrier. This project will reveal if tested materials are presented with promising profile upon using as direct pulp capping dressing in mechanical and carious-exposed pulp.

ELIGIBILITY:
Inclusion Criteria:

1. carious teeth that had no previous root canal treatment
2. Pulpal diagnosis of normal or reversible pulpitis

Exclusion Criteria:

1. History of irreversible pulpal pain
2. Immature teeth
3. Non restorable teeth
4. Teeth with active periodontal disease
5. History of any systemic disease
6. Concurrent medication with systemic steroids, antibiotics, analgesics, immunomodulatory drugs or cytotoxics

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
clinical vital pulp therapy success | from date of randomization until failure reported for up to 100 months
  Treatment was considered successful based on the absence of symptoms and signs Treatment was considered successful based on absence of symptoms and signs

SECONDARY OUTCOMES:
Radiographic success | from date of randomization until failure reported for up to 100 months
  treatment could be further evaluated based on the absence of canal oblitration

CONTACTS AND LOCATIONS:
Overall Officials: Lama Awawdeh, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Dental health center, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided